CLINICAL TRIAL: NCT01953796
Title: Study of Stair-step Clomiphene Protocol for Ovulation Induction in Women With Polycystic Ovarian Syndrome (PCOS) Compared to Traditional Protocol.
Brief Title: Clomiphene Stair-Step Protocol for Ovulation Induction in Women With Polycystic Ovarian Syndrome
Acronym: PCOSCCTvUSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kufa University (Other)
Responsible Party: Principal Investigator, Basima Shamkhi Al-Ghazali, Kufa university- Iraq, Kufa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kufa university
Record Dates: First submitted 2013-09-25; First posted 2013-10-01 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovarian Syndrome stair step traditional protocol
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study of Stair-step Clomiphene Protocol (Experimental): 50 mg clomiphene given for 5 days beginning on day 2 of the cycle. Tv USS done at days 11-14. When there is no response (no follicle >10 mm), 100 mg clomiphene is initiated immediately for 5 days, and U/S is repeated 1 week after the first tvUSS at day 21. If there is no response, another 150 mg clomiphene is initiated immediately for 5 days and U/S is performed 1week after the second U/S (day28). Ovulation for the stair-step cycles was confirmed by folliculometry (follicle tracing) by tvUSS.
  Interventions: Drug: clomiphene
- Traditional Protocol. (Active Comparator): Clomiphene medication was initiated at day two of the cycle. The starting dose was 50 mg/day for 5 consecutive days. In case of absent response, the patient was treated with 10 mg medroxyprogesterone acetate (MPA) for10 days. Daily doses of clomiphene citrate were increased by 50 mg in the next cycle up to 3 treatment cycle. In each cycle monitoring of follicular growth was done by tvUSS at day 11-14 of each cycle. First ovulation was used as the endpoint and the duration of follow-up was three treatment cycles (up to 150mg). Ovulation was assessed by tvUSS monitoring of follicle growth.
  Interventions: Drug: clomiphene

INTERVENTIONS:
Drug: clomiphene — For both protocols follow up of the follicular growth has been made by frequent tvUSS monitoring, which have the advantage of providing direct information about the size and number of follicle and measurement of endometrial thickness during clomiphene medication.
  Other Names: clomid

SUMMARY:
The objective of our study is to evaluate the efficacy of the clomiphene stair-step protocol to induce ovulation in women with polycystic ovarian syndrome (PCOS) compared to traditional protocol.

Methods:This was a randomized controlled clinical trial at the Fertility clinic of Al sadder teaching hospital at Al- Najaf city, Iraq . It included 140 women who met all of the inclusion criteria, they were divided into two groups; 65 patients for the stair step protocol and 75 patients for the traditional protocol.

DETAILED DESCRIPTION:
Overall study design This was a randomized clinical trial using toss a coin as randomization technique carried out on subfertile women attending the Fertility Clinic of AL Sadder Teaching Hospital at Al- Najaf city, Iraq from May 2010 till May 2011. 170 infertile women were selected at that time for study participation after their written consent.

Participant, recruitment and randomization:

The diagnostic criteria adopted for PCOS was according to Rotterdam ESHRE/ASRM sponsored PCOS consensus workshop group, 2004 based on the presence of two of the following three criteria: i.e. Oligo- and/or anovulation, hyperandrogenism clinical and/or biochemical, Polycystic ovaries, an ovary with 12 or more follicles measuring 2-9 mm indiameter and increased ovarian volume (>10 cm3) on transvaginal ultrasound(1) .

ELIGIBILITY:
Inclusion Criteria:Female in the reproductive age who is subfertile with the diagnosis of polycystic ovarian syndrome, serum FSH≤10 mIU/ml with spontaneous menses or positive bleeding response to progestagen withdrawal.

-

Exclusion Criteria:Male factor (moderate to severe) infertility, bilateral tubal blockage diagnosed by hystrosalpingographgy or laparoscopy and patients on metformin or other medication.

-

Ages: 21 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2010-05; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The time to ovulation with the stair step protocol was 21-28 days as compared with the traditional protocol which was 42 -70 days. | one year
  140 patients who met all of the inclusion criteria were divided into two main groups, Induction of ovulation for both protocols was performed.

CONTACTS AND LOCATIONS:
Overall Officials: basima sh jabbar, consultant, Principal Investigator — medical college/ kufa university
Locations (1):
- Basima Al- Ghazali, Najaf, Kufa, Iraq

REFERENCES:
- [Background] clomiphene protocol in polycystic ovarian syndrome: Hurst et al.
- [Result] Hurst BS, Hickman JM, Matthews ML, Usadi RS, Marshburn PB. Novel clomiphene "stair-step" protocol reduces time to ovulation in women with polycystic ovarian syndrome. Am J Obstet Gynecol. 2009 May;200(5):510.e1-4. doi: 10.1016/j.ajog.2008.10.031. Epub 2008 Dec 27. PMID 19114272